CLINICAL TRIAL: NCT06585215
Title: Expert Survey, Interactive Case Planning, and Modified Delphi Consensus: A Comprehensive Approach to Define Standards for Physician-Modified Stent Grafts in the Treatment of Abdominal Aortic Aneurysms
Brief Title: Standardization of Physician-Modified Stent Grafts for Abdominal Aortic Aneurysms
Acronym: RESTORE
Status: Enrolling by invitation | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Prouse Giorgio, MD, Ente Ospedaliero Cantonale, Bellinzona
Other Study IDs: ORLVasc-24-06
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Abdominal Aortic Aneurysm; Endovascular Procedures; Stents; Vascular Surgical Procedures
Keywords: EVAR; endovascular aneurysm repair; emergency aneurysm repair; AAA; abdominal aortic aneurysm; 3D printed graft; PMSG; PMSGs; physician-modified stent graft; custom fenestrated endografts; off-the-shelf branched devices; off-label endovascular devices; complex aneurysm management; parallel graft techniques; standardization in PMSG; procedural standardization in PMSG; PMEG; PMEGs; physician-modified endograft; 3D printing in medical applications
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study explores the use of physician-modified stent grafts (PMSGs) for treating abdominal aortic aneurysms that are unsuitable for open surgery or standard endovascular grafts. Custom-made fenestrated endografts are not viable in urgent or symptomatic cases due to lengthy manufacturing times. Although off-the-shelf branched devices are more readily available, they present challenges such as high costs, extensive thoracic coverage, limited long-term data, and anatomical restrictions. Parallel graft techniques are also associated with concerns regarding their durability. PMSG procedures, however, are not standardized and rely heavily on the physician's experience and expertise. The aim of this comprehensive study is to establish expert consensus on the indications, planning protocols, and procedural techniques for PMSGs.

DETAILED DESCRIPTION:
Principal Investigator: Dr. med. Giorgio Prouse

Ethics: The study was presented to the Ethics Committee of Canton Ticino, where formal approval was waived.

Background Physician-modified stent grafts (PMSGs) are increasingly used to treat urgent cases of symptomatic abdominal aortic aneurysms that are unfit for open surgery and cannot be treated with a standard endovascular graft. In symptomatic patients, custom-made fenestrated endografts are not an option due to the manufacturing time required. Recently, some off-the-shelf branched devices that allow for the treatment of many aneurysms involving the visceral aorta have been made available. However, these devices have significant shortcomings, including high cost, the need for extended thoracic aortic coverage, limited long-term outcome data, and the inability to treat certain anatomies. Parallel graft techniques have also been used for treating complex and urgent cases, yet the effectiveness and durability of aneurysm exclusion remain concerns. In such scenarios, PMSGs serve as a legitimate off-label alternative. However, the variety of techniques and strategies outlined by multiple study groups underscores the critical necessity for procedural standardization to mitigate the potential risks of life-threatening procedural errors.

Objective The study aims to establish a foundation for defining standards for PMSG procedures, including indications, optimal planning protocols, and the most established procedural techniques.

Primary Endpoint: To achieve expert consensus on aspects regarding indications, planning, and performing PMSGs in the treatment of abdominal aortic aneurysms, as determined by the completion of a modified Delphi consensus.

Secondary Endpoints:

* To conduct a survey-based scoping review to identify the predominant strategies and techniques utilized in the execution of PMSGs for interventions on abdominal aortic aneurysms.
* To test the hypothesis that 3D-printed models offer an advantage in terms of fenestration precision compared to CT-based planning methods.

Project Design and Procedures The project will consist of three separate sequential phases.

1. Phase: Global Cross-Sectional Survey Objective: To gather valuable real-world insights into the timing and methodology of PMSG procedures from vascular surgeons and interventional radiologists with expertise in fenestrated, branched, and PMSGs.

   Procedure:
   * Survey Design: A global cross-sectional survey consisting of 31 multiple-choice questions will be administered, focusing on indications for treatment, planning methodologies, and technical aspects of PMSG implementation.
   * Survey Platform: The survey will be built on the EDDDIE (Event Driven Direct Data Input Engine) platform hosted on the EOC server.
   * Participant Recruitment: A mailing list of vascular surgeons worldwide, sourced from published articles on PMSGs, will be used. Additionally, dedicated educational platforms and social media will support diffusion.
   * Survey Distribution: Emails will be sent containing a brief introductory page and a link to access the survey. The emails will be sent using an authenticated mail system by the EOC.

   Outcome: The survey will collect comprehensive data on the current practices and experiences of vascular surgeons in the field, providing insights into the timing, planning, and technical execution of PMSG procedures.
2. Phase: Case Planning Experiment Objective: To test the hypothesis that 3-D printed models offer an advantage in terms of fenestration precision compared to CT based planning methods. To this purpose this phase will involve a case planning experiment where participants from the survey will engage in planning a patient-specific PMSGs for two cases. These plannings will be compared with PMSGs created using 3D-printed templates of the two cases.

   Procedure:
   * Data Handling: Angio-CT scans from two patients treated for juxtarenal aneurysm with commercial fenestrated endografts will be anonymized and uploaded to a platform hosted on the EOC server.
   * Patient Consent: Both patients have signed informed consent for the re-utilization of clinical data for research purposes.
   * Platform and Software: The software used for image sharing is internal to EOC, with servers housed within the EOC structure. The system has been validated and complies with FDA CFR 21 Part 11 regulations.
   * Selection of Aortic Endografts: Four aortic endografts (one Medtronic Valiant Captivia Thoracic and one Medtronic Endurant II bifurcated for each patient) will be selected based on aortic diameter, with 20-30% oversizing.
   * 3D Model Generation: The CT scans of the patients will be loaded onto IntelliSpace Portal to generate .STL files. A lumen-based digital reconstruction will be performed with a 2 mm wall added. Patient-specific rigid 3D-printed aortic lumen templates will be produced for both patients using a Formalab 3B+ printer and transparent dental resin.
   * Production of Control PMSGs: The thoracic and abdominal grafts will be deployed inside the 3D templates, leaving a 2 cm sealing zone. The center of the fenestrations will be marked, and the diameter of the four visceral fenestrations measured. Fenestrations will be created using cautery and reinforced with a tip from a Cook Lunderquist guidewire sutured with 5-0 Prolene running suture.
   * Digital Mapping: The four fenestrated grafts will be mounted on an inner support and scanned to produce a digital 2D map of the graft. Anonymized angio-CT images will be uploaded to the sharing platform linked to the EDDDIE platform along with the corresponding digital 2D map of the grafts after digitally deleting the performed fenestrations.
   * Participant Involvement: Participants will choose their preferred device and perform planning of a PMSG for the two cases using their preferred imaging software. They will determine and draw the position and size of the fenestrations on the 2D map of the selected graft. Each fenestration map will be overlapped with the template fenestrated graft map to determine the difference in fenestration positions.

   Outcome Measures:
   * Position of the central point of the fenestration (angle degrees and distance from the proximal margin of stent fabric).
   * Diameter difference and percentage of surface overlap between corresponding fenestrations.

   Data Analysis: Outcome measures will be collected in a database and analyzed using statistical methods as described in the section.
3. Phase: Delphi Consensus Study (CREDES Guidelines) Objective: To establish a consensus on the issues identified as most critical in the survey of the first study phase and on the results from the comparative planning study.

Procedure:

* Panel Selection: Recruitment of experts in vascular surgery with extensive experience in PMSGs selected by the number of publications. Additionally, physicians known for their expertise in the field will be invited independently of the number of publications.
* Round 1: Panelists will review and rate statements and unresolved questions emerging from the cross-sectional survey and interactive planning analysis. They will provide ratings and may also explain choices with open text. Answers will be kept anonymous.
* Round 2: Feedback and Re-Assessment: A summary of the Round 1 results will be shared with panelists, highlighting areas of consensus and disagreement. Panelists will be able to reconsider their ratings in light of the group's feedback and provide justifications for their ratings. If necessary, a virtual meeting to clarify areas of disagreement may take place.
* Round 3: Final Consensus: Another summary of the Round 2 results will be shared. Panelists will re-rate the items, aiming for final consensus.

Consensus Definitions (Likert scale 1-5):

* Very high consensus: median = 5 and percentage agreement ≥ 80% IQR = 0
* High consensus: median = 4/5 percentage agreement ≥ 80% IQR = 0
* Moderate consensus: median ≥ 4; 60%-79% agreement IQR = 1
* Low consensus: median rating < 4 <60% agreement IQR > 1 Consensus Reporting: A final report will be provided with the panel's recommendations.

Outcome: The modified Delphi study will identify areas of strong consensus among experts, guiding best practices and standardizing PMSG procedures.

ELIGIBILITY:
Inclusion Criteria:

* Vascular Surgeons or Interventional Radiologists
* Must have expertise in fenestrated, branched, and PMSG procedures.
* Completed the 31-question survey via the EDDDIE platform.
* Informed consent is required for participation.

Exclusion Criteria:

* Physicians with no complex endovascular repair experience

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of vascular surgeons and interventional radiologists with specialized expertise in Physician-Modified Stent Grafts (PMSGs), fenestrated, or branched endografts. This population will include professionals with expertise in fenestrated, branched, and PMSGs. The survey aims to capture a global perspective, ensuring diverse representation from various healthcare systems. Participants must be willing to complete the survey online and provide informed consent to contribute their insights to this research.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06-14 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Expert Consensus on PMSG Indications and Techniques | 30.06.2025
  The expert consensus will be reached using the Delphi method (following CREDES guidelines), with three rounds planned. Consensus will be defined based on a Likert scale (1-5):
  * Very high consensus: median = 5 and percentage agreement ≥ 80%, IQR = 0;
  * High consensus: median = 4/5, percentage agreement ≥ 80%, IQR = 0;
  * Moderate consensus: median ≥ 4; 60%-79% agreement, IQR = 1;
  * Low consensus: median rating < 4, <60% agreement, IQR > 1

SECONDARY OUTCOMES:
Survey-Based Review of PMSG Strategies and Techniques | 30.06.2025
  * A global cross-sectional survey consisting of 31 multiple-choice questions will be administered.
  * Questions will use a mix of radio buttons and checkboxes to investigate three key areas: Indications for treatment, Planning methodologies, Technical aspects of PMSG implementation.
  * Survey responses will be analyzed to determine frequencies and percentages. We will also perform reliability analysis, inferential statistics, multivariate analysis, and qualitative analysis.
Comparison of 3D-Printed Models and CT-Based Planning | 30.06.2025
  * Participants from the survey will engage in planning a patient-specific PMSGs for two cases. These plannings will be compared with PMSGs created using 3D-printed templates of the two cases.
  * We will measure the position of the central point of the fenestration (angle degrees and distance from the proximal margin of stent fabric) and the diameter difference and percentage of surface overlap between corresponding fenestrations.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Prouse, Dr. med., Principal Investigator — Centro Vascolare Ticino
Locations (1):
- Centro Vascolare Ticino, Servizio di Chirurgia Vascolare e Angiologia, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Background] Rynio P, Gutowski P, Kazimierczak A. Physician-Modified Stent-Grafts Created in the Three-Dimensionally Aortic Template Have Better Reliability and Greater Alignment With the Target Vessels Than Stent-Grafts Modified Based on Measurements From Computed Tomography. J Endovasc Ther. 2023 Oct;30(5):769-778. doi: 10.1177/15266028221095396. Epub 2022 May 11. PMID 35543452
- [Background] Bortman J, Mahmood F, Schermerhorn M, Lo R, Swerdlow N, Mahmood F, Matyal R. Use of 3-Dimensional Printing to Create Patient-Specific Abdominal Aortic Aneurysm Models for Preoperative Planning. J Cardiothorac Vasc Anesth. 2019 May;33(5):1442-1446. doi: 10.1053/j.jvca.2018.08.011. Epub 2018 Aug 9. PMID 30217582
- [Background] Canonge J, Jayet J, Heim F, Chakfe N, Coggia M, Coscas R, Cochennec F. Comprehensive Review of Physician Modified Aortic Stent Grafts: Technical and Clinical Outcomes. Eur J Vasc Endovasc Surg. 2021 Apr;61(4):560-569. doi: 10.1016/j.ejvs.2021.01.019. Epub 2021 Feb 13. PMID 33589325
- [Background] Mitsuoka H, Terai Y, Miyano Y, Naitou T, Tanai J, Kawaguchi S, Goto S, Miura Y, Nakai M, Yamazaki F. Preoperative Planning for Physician-Modified Endografts Using a Three-Dimensional Printer. Ann Vasc Dis. 2019 Sep 25;12(3):334-339. doi: 10.3400/avd.ra.19-00062. PMID 31636743
- [Background] Georgiadis GS, van Herwaarden JA, Antoniou GA, Giannoukas AD, Lazarides MK, Moll FL. Fenestrated stent grafts for the treatment of complex aortic aneurysm disease: A mature treatment paradigm. Vasc Med. 2016 Jun;21(3):223-38. doi: 10.1177/1358863X16631841. Epub 2016 Mar 24. PMID 27013644
- [Background] Rynio P, Jedrzejczak T, Rybicka A, Milner R, Gutowski P, Kazimierczak A. Initial Experience with Fenestrated Physician-Modified Stent Grafts Using 3D Aortic Templates. J Clin Med. 2022 Apr 13;11(8):2180. doi: 10.3390/jcm11082180. PMID 35456273
- [Background] Haulon S, Barilla D, Tyrrell M, Tsilimparis N, Ricotta JJ 2nd. Debate: whether fenestrated endografts should be limited to a small number of specialized centers. J Vasc Surg. 2013 Mar;57(3):875-82. doi: 10.1016/j.jvs.2013.01.001. PMID 23446130
- [Background] Junger S, Payne SA, Brine J, Radbruch L, Brearley SG. Guidance on Conducting and REporting DElphi Studies (CREDES) in palliative care: Recommendations based on a methodological systematic review. Palliat Med. 2017 Sep;31(8):684-706. doi: 10.1177/0269216317690685. Epub 2017 Feb 13. PMID 28190381
- [Background] Nasa P, Jain R, Juneja D. Delphi methodology in healthcare research: How to decide its appropriateness. World J Methodol. 2021 Jul 20;11(4):116-129. doi: 10.5662/wjm.v11.i4.116. eCollection 2021 Jul 20. PMID 34322364

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT06585215/SAP_000.pdf